CLINICAL TRIAL: NCT00811759
Title: Open-label, Single Center, Uncontrolled Phase I/II Study Evaluating the Safety and Maximum Tolerated Dose of Daily Sorafenib Administered in Combination With Prolonged Temozolomide in Patients With Metastatic Melanoma
Brief Title: Sorafenib and Temozolomide in Treating Patients With Stage III or Stage IV Melanoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000626803; IGR-CSET-2006/1261; IGR-SORAF-TEM ST1; INCA-RECF0818; EUDRACT-2007-00527-18; SCHER-IGR-CSET-2006/1261; BAYER-IGR-CSET-2006/1261
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2009-07

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; stage III melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Sorafenib; Temozolomide; Gene Expression Profiling; Biopsy

INTERVENTIONS:
Drug: sorafenib tosylate
Drug: temozolomide
Genetic: gene expression analysis
Genetic: mutation analysis
Other: laboratory biomarker analysis
Other: pharmacological study
Procedure: biopsy

SUMMARY:
RATIONALE: Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving sorafenib together with temozolomide may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of giving sorafenib together with temozolomide in treating patients with stage III or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety profile and the maximum tolerated dose of sorafenib tosylate and temozolomide in patients with stage III-IV melanoma. (Phase I)
* Evaluate progression-free survival at 12 weeks. (Phase II)

Secondary

* Evaluate tumor response according to RECIST criteria.
* Evaluate overall and progression-free survival.
* Evaluate the effect of treatment on tumor vascularization.
* Compare the pharmacokinetic profile of temozolomide with and without sorafenib tosylate.
* Evaluate the number and the role of lymphocytes.
* Correlate tumor response rate with BRAF mutation status.
* Correlate response rate with MGMT activity.
* Compare the efficacy of genomics and proteomics as a means of discovery of serum biomarkers.
* Study the prognostic and predictive value of circulating endothelial cells and circulating endothelial progenitors.

OUTLINE: This is a phase I dose-escalation study followed by a phase II study.

Patients receive oral sorafenib tosylate twice daily on days 1-28 (days 8-28 of course 1) and oral temozolomide once daily on days 1-7 and 15-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients with accessible tumors (cutaneous or sub-cutaneous) undergo biopsies at baseline and day 28 for analysis of BRAF mutations and MGMT expression.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of unresectable or metastatic melanoma

  * Stage III or IV disease
* Previously treated or untreated metastatic disease
* At least one unidimensionally measurable lesion by RECIST criteria by scan or MRI
* No concurrent brain or CNS metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Life expectancy ≥ 3 months
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin > 9 g/dL
* PT, INR, and PTT < 1.5 times upper limit of normal (ULN)
* Transaminases < 2.5 times ULN (< 5 in the case of liver metastases)
* Amylase and lipase < 1.5 times ULN
* Bilirubin ≤ 1.5 times ULN
* Serum creatinine < 1.5 times ULN
* Normal respiratory, cardiac, and neurological function
* Not pregnant or nursing
* No history of any of the following cardiac conditions:

  * NYHA class II-IV heart failure
  * Coronary disease
  * Myocardial infarction within the past 6 months
  * Cardiac arrhythmia requiring treatment with something other than beta-blockers or digoxin
  * Severe uncontrolled hypertension
* No severe active infection > grade 2
* No epilepsy requiring medical treatment
* No other cancer except for carcinoma in situ of the cervix, basal cell carcinoma, superficial bladder tumors, or curatively treated cancer > 3 years ago
* No HIV or hepatitis B or C positivity
* No lactase or galactokinase deficiency, galactose intolerance, or disease accompanied by malabsorption of glucose or galactose
* No allergy to the study drugs or to dacarbazine
* Able to swallow medications
* No patients deprived of liberty
* No psychological, familial, social, or geographic conditions that would preclude clinical follow up

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior organ transplantation
* No prior temozolomide or sorafenib tosylate
* More than 30 days since other prior antitumor chemotherapy, immunotherapy, hormonal therapy, or investigational agent
* More than 30 days since prior study drugs
* More than 3 weeks since prior radiotherapy
* More than 3 weeks since prior biological response modifiers (i.e., filgrastim [G-CSF])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2007-06; Primary Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (Phase I)
Progression-free survival at 12 weeks (Phase II)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Robert, MD — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France